CLINICAL TRIAL: NCT00004223
Title: Phase II Trial of Gemcitabine and Docetaxel in Advanced Carcinoma of the Urothelium
Brief Title: Docetaxel and Gemcitabine in Treating Patients With Progressive Regional or Metastatic Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Treatment
Other Study IDs: CDR0000067464; E-2899
Record Dates: First submitted 2000-01-28; First posted 2004-02-25 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; posterior urethral cancer; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of docetaxel and gemcitabine in treating patients who have progressive regional or metastatic bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with progressive regional or metastatic transitional cell carcinoma of the urothelium and failure of only 1 prior systemic regimen treated with docetaxel and gemcitabine. II. Determine the toxicities of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive docetaxel IV over 1 hour followed by gemcitabine IV over 30 minutes on days 1 and 8. For patients with complete or partial response or stable disease at 3 weeks, treatment repeats every 3 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months through year 2, every 6 months through year 5, and then annually thereafter until disease progression.

PROJECTED ACCRUAL: A total of 22-45 patients will be accrued for this study over 18-21 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven progressive regional or metastatic transitional cell carcinoma of the urothelium or mixed histology containing a component of transitional cell carcinoma Failure of only 1 prior chemotherapy regimen for metastatic disease or in the adjuvant or neoadjuvant setting (not containing taxane or gemcitabine) Bidimensionally measurable disease No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 75,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 2.5 times upper limit of normal (ULN) if alkaline phosphatase normal OR Alkaline phosphatase no greater than 4 times ULN if SGOT normal OR SGOT less than 1.5 times ULN AND alkaline phosphatase less than 2.5 times ULN Renal: Creatinine no greater than 1.8 mg/dL Cardiovascular: No American Heart Association class III or IV heart disease No uncontrolled congestive heart failure No severe cardiac arrhythmias Neurologic: No sensory neuropathy grade 3 or 4 No prior peripheral neuropathy grade 2 or worse Other: No active unresolved infection being treated with parenteral antibiotics within the past 7 days No other malignancy within the past 5 years except: Curatively treated basal or squamous cell skin cancer or carcinoma in situ of the cervix Clinically unsuspected, organ confined prostate cancer found during cystoprostatectomy Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior systemic biologic response modifier therapy Prior intravesical BCG allowed Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 4 weeks since prior major surgery and recovered

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02-24 (Actual); Primary Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreicer, MD, FACP, Study Chair — The Cleveland Clinic
Locations (76):
- United States (73):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Kimball Medical Center, Lakewood, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Riverview Medical Center - Booker Cancer Center, Red Bank, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Result] Dreicer R, Manola J, Schneider DJ, Schwerkoske JF, George CS, Roth BJ, Wilding G; Eastern Cooperative Oncology Group. Phase II trial of gemcitabine and docetaxel in patients with advanced carcinoma of the urothelium: a trial of the Eastern Cooperative Oncology Group. Cancer. 2003 Jun 1;97(11):2743-7. doi: 10.1002/cncr.11413. PMID 12767086
- [Result] Manola JB, Dreicer R, Wilding G, et al.: Gemcitabine and docetaxel in advanced carcinoma of the urothelium: report of a phase II Eastern Cooperative Oncology Group trial . [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-796, 2002.